CLINICAL TRIAL: NCT01650012
Title: Pilot Trial of Hemodialysis Patient Aldosterone antagoniSm With Eplerenone Trial
Brief Title: Eplerenone in Hemodialysis Trial
Acronym: PHASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHASE-1
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Hemodialysis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eplerenone (Experimental): Target of 50 mg/day
  Interventions: Drug: eplerenone
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eplerenone — target 50 mg per day titrated down for hyperkalemia or hypotension
  Arms: Eplerenone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Forty percent of patients that require dialysis for kidney failure die within three years mostly due to heart disease. Heart failure and high blood pressure are common problems in patients that require dialysis and are key causes of death due to heart disease. Eplerenone is a drug that is very effective at improving heart failure and reducing blood pressure in patients that do not require dialysis. There is currently no evidence to tell physicians whether eplerenone would have similar benefits in patients that require dialysis. This evidence can only be reliably generated by performing a large scale study. Before such a study is undertaken, the investigators must determine whether eplerenone will be well tolerated and safe in patients that require dialysis. The investigators will perform an initial small trial called the Pilot trial in Hemodialysis patients undergoing Aldosterone antagoniSm with Eplerenone (PHASE) to determine if eplerenone is a well tolerated, safe medication to use in a very large, global study that will show whether or not eplerenone reduces important outcomes for patients like death from heart causes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* On hemodialysis >90 days
* Prescribed target body weight within 1 kg of current for all dialysis sessions within 4 weeks prior to randomization
* Able to provide written informed consent to participate

Exclusion Criteria:

* Occurrence of documented clinically important hypotension (systolic blood pressure <90 that required treatment) within 4 weeks of randomization
* Change in blood pressure medications within 4 weeks prior to randomization
* Occurrence of pre-dialysis serum potassium >6.0 mmol/L in 4 weeks prior to randomization
* Currently treated with and cannot withdraw spironolactone or eplerenone due to medical necessity
* Known allergy or sensitivity to eplerenone
* Pregnancy
* Scheduled living related donor renal transplant within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
permanent discontinuation of the study medication for hyperkalemia or permanent discontinuation of the study medication for hyperkalemia or hypotension | 13 weeks

SECONDARY OUTCOMES:
permanent discontinuation of study drug for any reason | 13 weeks
treatment adherence | 13 weeks
pre-dialysis potassium | 13 weeks
frequency of serious adverse events | 13 weeks
frequency of hospitalizations for a vascular reason | 13 weeks
fatal and non-fatal vascular events | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Walsh, Principal Investigator — McMaster University, Population Health Research Institute, St. Joseph's Hospital; Ron Wald, Principal Investigator — Keenan Research Centre, St. Michael's Hospital, University of Toronto
Locations (5):
- Canada (5):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138